CLINICAL TRIAL: NCT01237535
Title: Luteal Phase Support With Progesterone vs Estrogen and Progesterone on Pregnancy Rates in Ovarian Stimulation and Intrauterine Insemination Cycles: a Prospective Randomized Study
Brief Title: Luteal Phase Support With Progesterone Versus Estrogen and Progesterone on Pregnancy Rates
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Dr. Galia Oron, Rabin medical center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc005788ctil
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Unexplained Infertility; Mild Male Factor
Keywords: Unexplained infertility; Insemination; Luteal phase support; Ovarian stimulation
MeSH Terms: interventions — Estrogens; Progesterone; Insemination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Luteal support with progesterone only (Experimental): Luteal support with progesterone only (they will received vaginal P gel (Crinone 8% vaginal gel; Serono, Israel)Luteal support will begin after insemination and will be continued through the 12th week of gestation if the patient conceived.
  Interventions: Drug: Luteal support with progesterone only
- Luteal support with estrogen + progesterone (Experimental): Luteal support with estrogen + progesterone [(Crinone 8% vaginal gel; Serono, Israel) and Estrofem 4mg].
  Interventions: Drug: Luteal support with estrogen + progesterone
- No luteal support (No Intervention)
  Interventions: Procedure: Insemination without luteal support

INTERVENTIONS:
Drug: Luteal support with progesterone only — Luteal support with progesterone only (they will received vaginal P gel (Crinone 8% vaginal gel; Serono, Israel).Luteal support will begin after insemination and will be continued through the 12th week of gestation if the patient conceived.If no pregnancy will be achieved patients will undergo 3 treatment cycles preferably in the same treatment group.
  Arms: Luteal support with progesterone only
Drug: Luteal support with estrogen + progesterone — Luteal support with estrogen + progesterone [(Crinone 8% vaginal gel; Serono, Israel) and Estrofem 4mg].Luteal support will begin after insemination and will be continued through the 12th week of gestation if the patient conceived.If no pregnancy will be achieved patients will undergo 3 treatment cycles preferably in the same treatment group.
  Arms: Luteal support with estrogen + progesterone
Procedure: Insemination without luteal support — Routine insemination procedure without luteal support
  Arms: No luteal support

SUMMARY:
This is a single center, 3 arms, prospective randomized controlled open study to determine the impact of luteal phase support on pregnancy rates in ovarian stimulation and IUI cycles with recombinant FSH in patients with unexplained infertility and mild male factor.

Patients will be randomized into 3 groups:

1. Luteal support with progesterone only (they will received vaginal P gel (Crinone 8% vaginal gel; Serono, Israel)
2. Luteal support with estrogen + progesterone [(Crinone 8% vaginal gel; Serono, Israel) and Estrofem 4mg].
3. No luteal support

DETAILED DESCRIPTION:
Study design:

single center, 3 arms, prospective randomized controlled open study

Objective:

to determine the impact of luteal phase support on pregnancy rates in ovarian stimulation and IUI cycles with recombinant FSH in patients with unexplained infertility and mild male factor.

Methods:

All patients in all study groups will undergo a single insemination procedure and then will be randomized into 3 groups:

1. Luteal support with progesterone only (they will received vaginal P gel (Crinone 8% vaginal gel; Serono, Israel)
2. Luteal support with estrogen + progesterone [(Crinone 8% vaginal gel; Serono, Israel) and Estrofem 4mg].
3. No luteal support

Luteal support will begin after insemination and will be continued through the 12th week of gestation if the patient conceived. A pregnancy test will be performed 2 weeks after insemination (Serum hCG) an intrauterine pregnancy will be confirmed using a transvaginal ultrasound 2 weeks after a positive pregnancy test. If no pregnancy will be achieved patients will undergo 3 treatment cycles preferably in the same treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Couples with diagnosis of unexplained infertility
2. In their treatment cycle with ovarian stimulation and IUI using recombinant FSH in our institution.

Exclusion Criteria:

1. female partners with one or more of the following:

   * previous ovarian surgery
   * one ovary
   * polycystic ovaries on ultrasound examination
   * other endocrine abnormalities (i.e., polycystic ovarian syndrome, thyroid disorders,hyperprolactinemia,6.hypogonadotropic hypogonadism)
   * past ovarian hyperstimulation or hyperstimulation during the study period
   * diminished ovarian reserve (basal FSH level >15 IU/mL)
   * age of >40 years
2. sever male factor < 5 million total motile sperm on the day of insemination.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy | 4 weeks after insemintation
  A pregnancy test will be performed 2 weeks after insemination (Serum hCG) an intrauterine pregnancy will be confirmed using a transvaginal ultrasound 2 weeks after a positive pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Galia Oron, Dr, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel